CLINICAL TRIAL: NCT01076387
Title: A Prospective, Randomized Trial Comparing Robotic and Open Radical Cystectomy
Brief Title: Randomized Trial Comparing Robotic and Open Radical Cystectomy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 10-016
Record Dates: First submitted 2010-02-24; First posted 2010-02-26 (Estimated); Last update posted 2020-03-16 (Actual); Status verified 2020-03

CONDITIONS: Bladder Cancer
Keywords: Bladder; Cystectomy; Robotic; Open Radical; 10-016
MeSH Terms: conditions — Urinary Bladder Neoplasms

ARMS (2):
- open radical cystectomy (Active Comparator): This is a prospective, randomized study designed to compare two techniques of radical cystectomy with PLND (open and robotic) for bladder cancer.
  Interventions: Procedure: open radical cystectomy
- robotic-assisted radical cystectomy (Active Comparator): This is a prospective, randomized study designed to compare two techniques of radical cystectomy with PLND (open and robotic) for bladder cancer.
  Interventions: Procedure: robotic-assisted radical cystectomy

INTERVENTIONS:
Procedure: open radical cystectomy — Open radical cystectomy, pelvic lymph node dissection and open urinary diversion.
  Arms: open radical cystectomy
Procedure: robotic-assisted radical cystectomy — Robotic radical cystectomy, pelvic lymph node dissection and open urinary diversion. Robotic radical cystectomy is routinely performed by robotically trained and experienced minimally invasive surgeons.
  Arms: robotic-assisted radical cystectomy

SUMMARY:
The purpose of this study is to determine if using robotic surgical technology during bladder cancer surgery helps to reduce complications during and after the surgery. The removal of the bladder and lymph nodes will be done by a robotic or by an open technique. It may be a Robotic-assisted Radical Cystectomy (RARC) and Pelvic Lymph Node Dissection. Or it may be an Open Radical Cystectomy (ORC) and Pelvic Lymph Node Dissection.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years.
* Scheduled for radical cystectomy at MSKCC

Exclusion Criteria:

* Prior pelvic or abdominal radiation therapy;
* Prior extensive open abdominal surgery, defined by the discretion of the attending surgeon
* Any clinical contraindication for Trendelenburg positioning

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 124 (Actual)
Dates: Start 2010-02 (Actual); Primary Completion 2020-03-12 (Actual); Study Completion 2020-03-12 (Actual)

PRIMARY OUTCOMES:
To compare surgical complications of robotic-assisted radical cystectomy and open radical cystectomy. | intraoperative and 90-day postoperative period

SECONDARY OUTCOMES:
To examine clinical and pathological outcomes of robotic-assisted radical cystectomy and open radical cystectomy. | 2 years
Intra-operative performance (surgical time, blood loss) | time from anesthesia induction to final skin closure
Pathologic findings, including the stage specific, soft tissue surgical margin rate and number of lymph nodes removed. | 1.5 years
Bladder cancer recurrence (local, upper tract and distant disease) | 2 years
complications grade 2-5 | 2 years
  A secondary analysis will be used to determine if the total burden of grade 2-5 complications in the robotic arm is different from the open arm.
complication grade 3-5 | 2 years
  Determine if there is a difference in either the number of patients with grade 3-5 complication or the total number of grade 3-5 complication in the two arms of the study.

CONTACTS AND LOCATIONS:
Overall Officials: Vincent Laudone, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

REFERENCES:
- [Derived] Bochner BH, Dalbagni G, Sjoberg DD, Silberstein J, Keren Paz GE, Donat SM, Coleman JA, Mathew S, Vickers A, Schnorr GC, Feuerstein MA, Rapkin B, Parra RO, Herr HW, Laudone VP. Comparing Open Radical Cystectomy and Robot-assisted Laparoscopic Radical Cystectomy: A Randomized Clinical Trial. Eur Urol. 2015 Jun;67(6):1042-1050. doi: 10.1016/j.eururo.2014.11.043. Epub 2014 Dec 8. PMID 25496767
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm